CLINICAL TRIAL: NCT01764113
Title: Effect of Mindful Eating on Body Mass Index and Cardiovascular Risk Markers in Obese Adolescents: A Pilot Randomized Clinical Trial
Brief Title: Effect of Mindful Eating on Body Mass Index in Obese Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Seema Kumar, Assistant Professor of Pediatrics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-004401
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Adolescent Obesity
Keywords: Obesity; Adolescence; Mindful Eating
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindful Eating (Experimental): Subjects and at least one of their parents will receive mindful eating based behavioral modification program
  Interventions: Behavioral: Mindful Eating
- Standard Dietary Couseling (Active Comparator): Subjects and their parents will receive standard nutritional counseling provided by a registered dietician
  Interventions: Behavioral: Standard dietary counselling

INTERVENTIONS:
Behavioral: Mindful Eating — Subjects and their parents will receive mindful eating based behavioral modification program over multiple sessions
  Arms: Mindful Eating
Behavioral: Standard dietary counselling
  Arms: Standard Dietary Couseling

SUMMARY:
This study is designed to study the effect of a family based mindfulness training program with special focus on diet and nutrition on weight and cardiovascular risk markers in obese adolescents.

DETAILED DESCRIPTION:
40 obese adolescents would be randomized into either a mindfulness based behavioral modification program or standard dietary counseling. At least one parent would be expected to attend the counseling sessions. Patients would be followed for a period of 6 months. Anthropometric parameters, questionaiires relating to quality of life and blood tests would be drawn at baseline and and at 6 months.

ELIGIBILITY:
Inclusion Criteria

* BMI at or greater than the 95th percentile for age and gender

Exclusion Criteria

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Baseline and 6 months
  Body Mass Index would be calculated at baseline, at 3 months and at 6 months

SECONDARY OUTCOMES:
Quality of Life | Baseline and 6 months
  Well validated questionnaires of quality of life would be assessed at baseline, at 3 months and at 6 months.

OTHER OUTCOMES:
Fasting glucose | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States